CLINICAL TRIAL: NCT00913536
Title: Cone-Beam Computed Tomography in Image-Guided Radiotherapy for Patients With Bladder Cancer
Brief Title: Cone Beam Computed Tomography (CT) Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 05-0620-CE
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Cone Beam CT; On-line image guidance; Radiation therapy in bladder cancer patients
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cone beam CT in Bladder Cancer (Experimental)
  Interventions: Other: Using Cone beam CT in patients with Bladder Cancer

INTERVENTIONS:
Other: Using Cone beam CT in patients with Bladder Cancer — Using cone beam CT scanner will help to increase the accuracy of your radiotherapy treatment. The cone beam CT scanner is a part of the radiotherapy treatment unit.

SUMMARY:
This study is designed to investigate whether daily images of the pelvis and bladder using a device called a cone beam CT scanner will help to increase the accuracy of radiotherapy treatment. The cone beam CT scanner is a part of the radiotherapy treatment unit. The results of the study may allow patients in the future who are undergoing radiotherapy treatment for bladder cancer to 1) have more accurately directed treatment, 2) have higher doses of radiation delivered to the tumour while keeping doses to the surrounding normal tissues as low as possible. This may allow eradication of the cancer while minimizing side effects of treatment.

This study consists of two phases: Phase A and Phase B. In Phase A, images were collected and analyzed and it was confirmed that it was useful to use the cone beam machine for daily Cone Beam CT Bladder (Phase B)treatment adjustments. In phase B, we hope to be able to use cone beam CT scans to more accurately direct the radiotherapy treatments on a daily basis.

DETAILED DESCRIPTION:
Cone beam computed tomography (CT) is new technology that allows the acquisition of 3-dimensional cross-sectional imaging while the patient is positioned on a linear accelerator couch. Cone beam CT also provides 3D soft tissue volumetric data and therefore important information on daily interfraction movement and deformation of normal critical structures within the pelvis. Visualization of the tumor using this technology may also be enhanced by the additional placement of fiducial markers around the tumor bed to ensure even more accurate targeting. The aim of this study is to assess the feasibility of daily cone beam CT for image guidance in patients receiving radiation therapy (RT) for bladder cancer as well document changes in size and location of the bladder and rectum during an entire course of RT. This will enable us to explore techniques for radiation therapy based on normal tissue avoidance models to reduce treatment toxicity and potentially dose escalation in the future.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of carcinoma of the bladder

* Patients undergoing radical external beam radiotherapy
* Age >18 years
* ECOG performance status 0-1
* Informed consent

Exclusion Criteria:

* Inflammatory bowel disease or collagen vascular disease
* Patients undergoing palliative radiotherapy to the bladder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-11 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of cone beam CT for daily on-line image guidance in patients receiving radiation therapy for bladder cancer. | 5 years

SECONDARY OUTCOMES:
Measure interfraction,intrafraction & deformity of bladder;determine adequacy of present margins; report bladder volume changes during treatment; evaluate use of fiducial markers plus CBCT for on-line image guidance & transabdominal ultrasound system. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Chung, MB ChB, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada